CLINICAL TRIAL: NCT03841786
Title: Effect of Phosphorus Additives on the Metabolome in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Orlando M. Gutierrez, MD, MMSc, Primary Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: IRB-300002442
Record Dates: First submitted 2019-02-12; First posted 2019-02-15 (Actual); Last update posted 2022-12-29 (Actual); Status verified 2022-12

CONDITIONS: Metabolic Syndrome; Insulin Sensitivity; Cardiovascular Diseases
Keywords: Metabolome; Phosphorus; Nutrition
MeSH Terms: conditions — Metabolic Syndrome; Insulin Resistance; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: Eligible subjects will consume a phosphorus supplemented diet (study diet) and a sodium and potassium chloride supplemented diet (control diet), with cross-over to the other diet following a 24-day wash-out period. The order in which the diets are consumed will be randomly assigned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control diet (Placebo Comparator): Participants will be asked to consume a normal diet supplemented with sodium chloride (sodium chloride tablets, USP, 1 gram; 3 tablets per day) and potassium chloride (Klor-Con, 8 mEq; 0.5 tablets per day) for 1 week.
  Interventions: Other: Control Diet
- Phosphorus-supplemented study diet (Experimental): Participants will be instructed to consume a normal diet with supplemental phosphorus (K-Phos Neutral tablets, 250 mg; 4 tablets a day) for 1 week.
  Interventions: Other: Phosphorus-supplemented study diet

INTERVENTIONS:
Other: Phosphorus-supplemented study diet — Participants will be instructed to consume a normal diet and will take a total of 1,000 mg of supplemental phosphorus per day in the form of neutral sodium phosphorus (K-Phos neutral®) for 1 week.
  Arms: Phosphorus-supplemented study diet
Other: Control Diet — Participants will be asked to consume a normal diet supplemented with sodium and potassium chloride tablets commensurate with the extra sodium and potassium content consumed during the study diet period for 1 week
  Arms: Control diet

SUMMARY:
This study evaluates the effect of phosphorus supplementation on the human metabolome. The investigators will do so by conducting a cross-over study in healthy adults consuming a study diet (normal diet supplemented by neutral sodium phosphorus, 1 gram/day) for seven days and a control diet (normal diet supplemented by sodium and potassium chloride only) for seven days with a 28 day wash-out period in between. Untargeted metabolomic analyses will be done in serum samples obtained at the end of each diet period.

DETAILED DESCRIPTION:
Phosphorus is an essential micronutrient involved in a number of key biological processes. Excess phosphorus intake is linked to hypertension, heart failure, and disorders of bone and mineral metabolism. This has critical implications for public health in that dietary phosphorus consumption in the US far exceeds current recommendations for daily intake.

Most studies that examined the adverse effects of excess phosphorus intake have focused on single tissue or cell specific processes. However, a full understanding of the systemic impact of nutritional phosphorus intake requires a more integrated biologic approach. The human metabolome represents the final end-product of the omics cascade, which can serve as an integrated measure of the total biological response to dietary exposures. Few studies have examined the impact of nutritional phosphorus intake on the human metabolome. Expanding the understanding of the effect of diet phosphorus on the metabolome has the potential to identify novel phosphorus-responsive pathways that may be therapeutic targets for reducing the development of hypertension, cardiovascular and kidney disease. The investigators will test the following hypothesis: consumption of a high phosphorus diet will result in significant changes in circulating metabolites associated with cardiometabolic health.

This hypothesis is supported by published and preliminary studies showing that high phosphorus intake alters metabolic pathways with a wide variety of pathophysiologic effects. In the current application, the investigators propose to build on this work by investigating the effect of phosphorus consumption on the human metabolome using an untargeted approach. The investigators will do so by conducting a cross-over study in healthy adults consuming a study diet (normal diet supplemented by neutral sodium phosphorus, 1 gram/day) for seven days and a control diet (normal diet supplemented by sodium and potassium chloride only) for seven days with a 28 day wash-out period.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers, aged 18 - 45 years with normal kidney function (estimated glomerular filtration rate > 60 ml/min/1.73m2).

Exclusion Criteria:

* abnormal urinalysis-presence of hematuria, proteinuria, or leukocyturia. pregnancy or breast-feeding
* Medical conditions impacting phosphate metabolism-primary hyperparathyroidism; gastrointestinal malabsorption disorders such as Crohn's Disease, ulcerative colitis, celiac disease, or liver dysfunction; hyper- or hypothyroidism; irregular menses for female subjects.
* Medications known to affect phosphorus metabolism- current use of phosphorus supplements, high-dose or activated vitamin D compounds, regular antacid or laxative use, anticonvulsants.
* Hyper- or hypophosphatemia (≥ 4.6 mg/dl or ≤ 2.5 mg/dl respectively), hyper- or hypocalcemia (≥ 10.6 or ≤ 8.5 mg/dl respectively), or severe anemia (hemoglobin < 8 g/dl for women and < 9 g/dl for men), hyperkalemia (potassium > 5.0 mmol/L).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-06-28 (Actual); Primary Completion 2021-04-27 (Actual); Study Completion 2022-09-15 (Actual)

PRIMARY OUTCOMES:
Untargeted Metabolomics | 7 days
  Untargeted metabolomics will be the primary endpoint and will be performed on serum samples obtained for all participants at the end of each dietary period.

SECONDARY OUTCOMES:
Fibroblast growth factor 23 (FGF23) | 7 days
  FGF23 concentrations will be measured at the end of each dietary period

CONTACTS AND LOCATIONS:
Overall Officials: Orlando Gutierrez, M.D., Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Block GA, Klassen PS, Lazarus JM, Ofsthun N, Lowrie EG, Chertow GM. Mineral metabolism, mortality, and morbidity in maintenance hemodialysis. J Am Soc Nephrol. 2004 Aug;15(8):2208-18. doi: 10.1097/01.ASN.0000133041.27682.A2. PMID 15284307
- [Background] Dhingra R, Sullivan LM, Fox CS, Wang TJ, D'Agostino RB Sr, Gaziano JM, Vasan RS. Relations of serum phosphorus and calcium levels to the incidence of cardiovascular disease in the community. Arch Intern Med. 2007 May 14;167(9):879-85. doi: 10.1001/archinte.167.9.879. PMID 17502528
- [Background] Foley RN, Collins AJ, Herzog CA, Ishani A, Kalra PA. Serum phosphate and left ventricular hypertrophy in young adults: the coronary artery risk development in young adults study. Kidney Blood Press Res. 2009;32(1):37-44. doi: 10.1159/000203348. Epub 2009 Feb 20. PMID 19229116
- [Background] Ix JH, De Boer IH, Peralta CA, Adeney KL, Duprez DA, Jenny NS, Siscovick DS, Kestenbaum BR. Serum phosphorus concentrations and arterial stiffness among individuals with normal kidney function to moderate kidney disease in MESA. Clin J Am Soc Nephrol. 2009 Mar;4(3):609-15. doi: 10.2215/CJN.04100808. Epub 2009 Feb 11. PMID 19211667
- [Background] Kestenbaum B, Sampson JN, Rudser KD, Patterson DJ, Seliger SL, Young B, Sherrard DJ, Andress DL. Serum phosphate levels and mortality risk among people with chronic kidney disease. J Am Soc Nephrol. 2005 Feb;16(2):520-8. doi: 10.1681/ASN.2004070602. Epub 2004 Dec 22. PMID 15615819
- [Background] Tonelli M, Sacks F, Pfeffer M, Gao Z, Curhan G; Cholesterol And Recurrent Events Trial Investigators. Relation between serum phosphate level and cardiovascular event rate in people with coronary disease. Circulation. 2005 Oct 25;112(17):2627-33. doi: 10.1161/CIRCULATIONAHA.105.553198. PMID 16246962
- [Background] Mathew S, Tustison KS, Sugatani T, Chaudhary LR, Rifas L, Hruska KA. The mechanism of phosphorus as a cardiovascular risk factor in CKD. J Am Soc Nephrol. 2008 Jun;19(6):1092-105. doi: 10.1681/ASN.2007070760. Epub 2008 Apr 16. PMID 18417722
- [Background] Shuto E, Taketani Y, Tanaka R, Harada N, Isshiki M, Sato M, Nashiki K, Amo K, Yamamoto H, Higashi Y, Nakaya Y, Takeda E. Dietary phosphorus acutely impairs endothelial function. J Am Soc Nephrol. 2009 Jul;20(7):1504-12. doi: 10.1681/ASN.2008101106. Epub 2009 Apr 30. PMID 19406976
- [Background] Adeney KL, Siscovick DS, Ix JH, Seliger SL, Shlipak MG, Jenny NS, Kestenbaum BR. Association of serum phosphate with vascular and valvular calcification in moderate CKD. J Am Soc Nephrol. 2009 Feb;20(2):381-7. doi: 10.1681/ASN.2008040349. Epub 2008 Dec 10. PMID 19073826
- [Background] Saab G, Whooley MA, Schiller NB, Ix JH. Association of serum phosphorus with left ventricular mass in men and women with stable cardiovascular disease: data from the Heart and Soul Study. Am J Kidney Dis. 2010 Sep;56(3):496-505. doi: 10.1053/j.ajkd.2010.03.030. Epub 2010 Jun 26. PMID 20580478
- [Background] Gutierrez OM. Fibroblast growth factor 23 and disordered vitamin D metabolism in chronic kidney disease: updating the "trade-off" hypothesis. Clin J Am Soc Nephrol. 2010 Sep;5(9):1710-6. doi: 10.2215/CJN.02640310. Epub 2010 May 27. PMID 20507957
- [Background] Uribarri J. Phosphorus homeostasis in normal health and in chronic kidney disease patients with special emphasis on dietary phosphorus intake. Semin Dial. 2007 Jul-Aug;20(4):295-301. doi: 10.1111/j.1525-139X.2007.00309.x. PMID 17635818
- [Background] Uribarri J, Calvo MS. Hidden sources of phosphorus in the typical American diet: does it matter in nephrology? Semin Dial. 2003 May-Jun;16(3):186-8. doi: 10.1046/j.1525-139x.2003.16037.x. PMID 12753675
- [Background] Gutierrez OM, Luzuriaga-McPherson A, Lin Y, Gilbert LC, Ha SW, Beck GR Jr. Impact of Phosphorus-Based Food Additives on Bone and Mineral Metabolism. J Clin Endocrinol Metab. 2015 Nov;100(11):4264-71. doi: 10.1210/jc.2015-2279. Epub 2015 Aug 31. PMID 26323022